CLINICAL TRIAL: NCT04829214
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study of OTO-313 Given as a Single Intratympanic Injection in Subjects With Unilateral Subjective Tinnitus
Brief Title: OTO-313 in Subjects With Unilateral Subjective Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OTO-313-201
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Subjective Tinnitus
Keywords: intratympanic injection; IT injection; gacyclidine; tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, multicenter
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTO-313 (Experimental)
  Interventions: Drug: OTO-313
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OTO-313 — Single intratympanic injection
  Arms: OTO-313
Drug: Placebo — Single intratympanic injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of OTO-313 in subjects with unilateral tinnitus and to determine the safety and tolerability of OTO-313 in subjects with unilateral tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Subject has early-onset subjective unilateral tinnitus that is persistent (consistently aware of their tinnitus throughout much of the waking day).
* Subject is able to use the diary to complete their daily tinnitus ratings.
* Subject's tinnitus is likely of cochlear origin, e.g., associated with sensorineural hearing loss; acute hearing loss from noise trauma, barotrauma, or traumatic cochlear injury (acute acoustic trauma, blast trauma, middle ear surgery, inner ear barotrauma); age related hearing loss; resolved otitis media; ototoxic drug exposure.
* Subject is willing to comply with the protocol and attend all study visits.

Exclusion Criteria:

* Subject has pulsatile tinnitus, temporomandibular joint disease (TMJ) associated with tinnitus perception, tinnitus resulting from traumatic head or neck injury, or tinnitus resulting from a tumor or stroke.
* Subject is pregnant, lactating, or undergoing fertility treatment.
* Subject has other clinically significant illness, medical condition or medical history at Screening or Baseline that, in the Investigator's opinion, would likely reduce the safety of study participation or compliance with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (31):
  - Central California Clinical Research, Fresno, California
  - Breathe Clear Institute, Torrance, California
  - University of Colorado, Department of Otolaryngology, Aurora, Colorado
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - ENT and Allergy Associates of FL, Boynton Beach, Florida
  - ENT and Allergy Associates of Florida, LLC, Delray Beach, Florida
  - Research Centers of America, Hollywood, Florida
  - ENT and Allergy Associates of Florida, LLC, Plantation, Florida
  - ENT and Allergy Associates of Florida, LLC, Port Saint Lucie, Florida
  - Ear Research Foundation, Sarasota, Florida
  - Rush University Medical Center, Chicago, Illinois
  - ChicagoENT, Chicago, Illinois
  - Kentuckian Ear, Nose & Throat, Louisville, Kentucky
  - Advanced ENT and Allergy, PLLC, Louisville, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Center for Specialized Medicine, Department of Otolaryngology-Head and Neck Surgery, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center/Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - Dent Neurosciences Research Center, Amherst, New York
  - Charlotte Eye Ear Nose & Throat Associates, P.A., Matthews, North Carolina
  - Piedmont Ear, Nose & Throat Associates, PA, Winston-Salem, North Carolina
  - UC Health Otolaryngology-Head and Neck Surgery, Cincinnati, Ohio
  - Department of Otolaryngology-Head and Neck Surgery, Medical University of South Carolina, Charleston, South Carolina
  - Carolina Ear, Nose & Throat Clinic/CENTRI Inc., Orangeburg, South Carolina
  - Spartanburg/Greer ENT & Allergy, Spartanburg, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Fort Worth ENT, Fort Worth, Texas
  - ENT Associates of Texas, McKinney, Texas
  - Alamo ENT Associates, San Antonio, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Eastern Virginia Medical School Department of Otolatyngology, Norfolk, Virginia
  - Advanced Otolaryngology, P.C. DBA Richmond ENT, Richmond, Virginia
- Germany (8):
  - HNO Praxis - Marianne Grohe, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - HNO - Praxis Göttingen, Göttingen
  - HNO Praxis am Necker, Heidelberg
  - HNO-Gemeinschaftspraxis, Heidelberg
  - Department of Otorhinolaryngology, Head and Neck Surgery, University Hospital, Jena
  - Universitätsklinikum Mannheim Klinik für Otorhinolaryngologie, Kopf- und Halschirurgie, Mannheim
  - Klinikum der Universitaet Muenchen, München
- Poland (4):
  - Centrum Medyczne Kwiatowa, Bydgoszcz
  - Centrum Medyczne ZDROWA, Krakow
  - Centrum Medyczne PROMED, Krakow
  - MT Medic Specjalistyczna Pralctyka Lekarska Tomasz Stapiński, Krosno
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - NHS Tayside, Dundee
  - University Hospitals of Leicester NHS Trust, Leicester
  - Norfolk and Norwich University Hospitals NHS Trust, Norwich
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 56 clinical centers were approved in Germany, Poland, United States, and United Kingdom to conduct this study. Thirty-six centers enrolled subjects. First subject was randomized 04 May 2021; Last subject was randomized 21 February 2022.
Pre-assignment Details: All subjects registered for this study signed an informed consent and entered a lead-in period. Following Lead-in, 153 subjects were randomized (=Full Analysis Set) and 151 subjects received study drug (=Safety Analysis Set). The most common reason for not being randomized was too low a score on the Tinnitus Functional Index (TFI)..
Groups:
- OTO-313: OTO-313: Single intratympanic 200 microliter injection of gacyclidine solution in medium chain triglycerides (0.16 mg/mL)
- Placebo: Placebo: Single intratympanic 200 microliter injection of medium chain triglycerides (OTO-313 vehicle)
Period: Randomization
Arm/Group | OTO-313 | Placebo
Started | 77 | 76
Completed | 77 | 76
Not Completed | 0 | 0
Period: Follow-up and Efficacy Analysis
Arm/Group | OTO-313 | Placebo
Started | 77 | 76
Completed | 70 | 72
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTO-313 | Placebo | Total
Number analyzed (Participants) | 77 | 76 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.75) | 50.8 (15.22) | 51.6 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 36 | 38 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 67 | 68 | 135
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 67 | 68 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 57 | 57 | 114
  Poland | 13 | 12 | 25
  United Kingdom | 1 | 0 | 1
  Germany | 6 | 7 | 13
Duration of Tinnitus [Count of Participants; unit: Participants]
  ≥2 to ≤6 months | 33 | 33 | 66
  >6 to ≤12 months | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Tinnitus Functional Index (TFI) Responders at Weeks 4 and at Week 8
Description: The TFI is a validated, 25-item questionnaire; index score from 0 to 100; higher scores indicate a greater problem with tinnitus. A responder is considered as any subject with at least a 13-point improvement from Baseline on the (TFI). This responder analysis required both Week 4 and Week 8 to have a 13-point improvement from Baseline.
Time Frame: Week 4 and Week 8 (both had to meet criterion for the subject to be considered a "responder")
Measure: Count of Participants; unit: Participants
Groups:
- OTO-313 Full Analysis Set: The OTO-313 full analysis set includes all subjects randomized to OTO-313 and analyzed in this group utilizing the intent-to-treat principle.
- Placebo Full Analysis Set: The placebo full analysis set includes all subjects randomized to placebo and analyzed in this group utilizing the intent-to-treat principle.
Arm/Group | OTO-313 Full Analysis Set | Placebo Full Analysis Set
Number analyzed (Participants) | 77 | 76
Participants | 20 | 27
Statistical Analysis 1: Comparison: OTO-313 Full Analysis Set vs Placebo Full Analysis Set; The percentage of responders will be compared between the two groups using the Mantel Haenszel test controlling for category of duration of tinnitus and category of baseline TFI overall score. The primary efficacy analysis will be conducted for the comparison of OTO-313 and placebo, using a 2-sided test and an alpha level of 5%. The 95% confidence intervals (CI) around the common risk difference will also be provided; Test type: Superiority; p = 0.385, Mantel Haenszel; Risk Difference (RD) = -10.2, 95% CI 2-sided [-26 to 5], Standard Error of Mean 7.9

2. Secondary Outcome: Change From Baseline in Daily Tinnitus Loudness at Week 8
Description: Numerical rating scale (NRS) from 0 (No Tinnitus) to 10 (Extremely Loud Tinnitus) collected every day. Post-baseline weekly NRS scores will be calculated as the average score of all recorded diary entries within each study week.
Time Frame: The average is calculated for the Baseline and for each study week. Reported here is the change from Baseline to Week 8.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTO-313 Full Analysis Set | Placebo Full Analysis Set
Number analyzed (Participants) | 77 | 76
units on a scale | -0.67 (1.767) | -0.90 (1.557)

3. Secondary Outcome: Change From Baseline in Daily Tinnitus Annoyance at Week 8
Description: Numerical rating scale from 0 (Not Annoying) to 10 (Extremely Annoying) collected every day. Post-baseline weekly NRS scores will be calculated as the average score of all recorded diary entries within each study week.
Time Frame: The average is calculated for the Baseline and for each study week. Reported here is the change from Baseline to Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OTO-313 Full Analysis Set | Placebo Full Analysis Set
Number analyzed (Participants) | 77 | 76
units on a scale | -0.73 (1.910) | -1.11 (1.804)

4. Secondary Outcome: Patient Global Impression of Change at Week 8
Description: Change in overall tinnitus status as perceived by the subject as assessed at the Week 8 visit. Subjects were asked, "Since the beginning of the clinical study, how would you rate your tinnitus?" and had the choice to answer from very much worse (-3) to very much improved (3). The mean change from baseline at Week 8 is reported here.
Time Frame: Week 8 reported here
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | OTO-313 Full Analysis Set | Placebo Full Analysis Set
Number analyzed (Participants) | 77 | 76
score on a scale | 0.32 (0.139) | 0.36 (0.138)

5. Other Pre Specified Outcome: Otoscopic Examinations - Presence of Perforation in the Treated Ear at Week 16 (Final Visit)
Description: Ear examinations were done at every visit. One of the important safety endpoints is an observation of a perforation in the ear drum that did not heal properly after the injection. Reported here are the Week 16 (final visit) results.
Time Frame: After dosing (Baseline) up to end of study (16 Weeks)
Measure: Count of Participants; unit: Participants
Groups:
- OTO-313 Safety Analysis Set: Subjects randomized to OTO-313 and received a dose of OTO-313.
- Placebo Safety Analysis Set: Subjects randomized to placebo and received placebo.
Arm/Group | OTO-313 Safety Analysis Set | Placebo Safety Analysis Set
Number analyzed (Participants) | 77 | 74
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded as observed or reported during or after dosing up to the final visit (Week 16).
Arm/Group | OTO-313 Safety Analysis Set | Placebo Safety Analysis Set
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/76
Serious Adverse Events (participants affected / at risk) | 2/77 | 0/76
Other Adverse Events (participants affected / at risk) | 23/77 | 24/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-313 Safety Analysis Set (N=77) | Placebo Safety Analysis Set (N=76)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTO-313 Safety Analysis Set (N=77) | Placebo Safety Analysis Set (N=76)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Blood Potassium Increased (Investigations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 8 (8) | 8 (8)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5) | 7 (7)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Viral Sinusitis (Infections and infestations) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT04829214/Prot_SAP_000.pdf